CLINICAL TRIAL: NCT04720183
Title: A Phase 1, Fixed Sequence, Open-label, Drug-drug Interaction Study to Evaluate the Effect of GLPG3970 on the Pharmacokinetics of Sulfasalazine in Adult, Healthy Subjects
Brief Title: Drug-drug Interaction Study with GLPG3970 and Sulfasalazine in Adult, Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: GLPG3970-CL-117
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-07

CONDITIONS: Healthy
MeSH Terms: interventions — Sulfasalazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sulfasalazine + GLPG3970 (Experimental)
  Interventions: Drug: Sulfasalazine; Drug: GLPG3970

INTERVENTIONS:
Drug: Sulfasalazine — On Day 1, Day 5 and Day 9, a single oral dose of sulfasalazine tablets in fasted state.
Drug: GLPG3970 — On Day 5 and Day 9, a single dose of GLPG3970 oral solution in fasted state.

SUMMARY:
GLPG3970 will be given with sulfasalazine to investigate the effect of co-administration on the pharmacokinetics of sulfasalazine, and on the safety and tolerability of the drugs in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age (extremes included), on the date of signing the informed consent form (ICF). Females should be of non-childbearing potential.
* A body mass index (BMI) between 18.0 to 30.0 kg/m2, inclusive.
* A breast cancer resistance protein (BCRP) c421C/C genotype.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and fasting clinical laboratory safety tests, available at screening and prior to the first sulfasalazine administration. Bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) must be no greater than 1.5x upper limit of normal range (ULN). Other clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered not clinically significant in the opinion of the investigator.

This list only contains the key inclusion criteria.

Exclusion Criteria:

* Known hypersensitivity to the investigational product (IP) (GLPG3970), or sulfasalazine, or sulfa drugs, or to their ingredients, or history of a significant allergic reaction to IP or sulfasalazine ingredients as determined by the investigator.
* Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) or history of hepatitis from any cause with the exception of hepatitis A that was resolved at least 3 months prior to first dosing of sulfasalazine.
* History of or a current immunosuppressive condition (e.g. human immunodeficiency virus (HIV) infection).
* Having any illness, judged by the investigator as clinically significant, in the 3 months prior to first dosing of sulfasalazine.
* Presence or sequelae of gastrointestinal, liver, kidney (estimated glomerular filtration rate (eGFR) <=90 mL/min/1.73 m2, using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula) or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Subjects with an N-acetyltransferase 2 (NAT2) slow acetylator genotype.

This list only contains the key exclusion criteria.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of sulfasalazine | Between Day 1 pre-dose and Day 12
  To evaluate the effect of GLPG3970 on the pharmacokinetics (PK) of sulfasalazine and its active metabolite sulfapyridine in healthy subjects.
Cmax of sulfapyridine | Between Day 1 pre-dose and Day 12
  To evaluate the effect of GLPG3970 on the pharmacokinetics (PK) of sulfasalazine and its active metabolite sulfapyridine in healthy subjects.
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) of sulfasalazine | Between Day 1 pre-dose and Day 12
  To evaluate the effect of GLPG3970 on the pharmacokinetics (PK) of sulfasalazine and its active metabolite sulfapyridine in healthy subjects.
AUC0-inf of sulfapyridine | Between Day 1 pre-dose and Day 12
  To evaluate the effect of GLPG3970 on the pharmacokinetics (PK) of sulfasalazine and its active metabolite sulfapyridine in healthy subjects.
Sulfapyridine to sulfasalazine AUC ratio | Between Day 1 pre-dose and Day 12
  To evaluate the effect of GLPG3970 on the pharmacokinetics (PK) of sulfasalazine and its active metabolite sulfapyridine in healthy subjects.

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) by Severity | From Day 1 through study completion, an average of 1 month
  To evaluate the safety and tolerability of the coadministration of GLPG3970 with sulfasalazine in healthy subjects
Maximum observed concentration (Cmax) of GLPG3970 | Between Day 5 pre-dose and Day 10
  To evaluate the PK of GLPG3970 in presence of sulfasalazine in healthy subjects
Area under the plasma concentration-time curve from time zero till the last observed quantifiable concentration (AUC0-t) | Between Day 5 pre-dose and Day 10
  To evaluate the PK of GLPG3970 in presence of sulfasalazine in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Rueda-Rincon, MD, Study Director — Galapagos NV
Locations (1):
- Biotral Inc, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No